CLINICAL TRIAL: NCT00801658
Title: Efficacy of SLT in Patients With Insufficient IOP Control Under Maximum Tolerated Drug Therapy (Eye Drops)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Ellex Medical Pty, 82 Gilbert Str., Adelaide, SA 5000 (Unknown)
Responsible Party: Prof. Dr. Dr. Jens Funk, University hospital zurich, eye clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FunkSLT
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Glaucoma
Keywords: glaucoma; SLT; Laser treatment; IOP; glaucoma treated with eye drops but IOP not controlled
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: selective Laser Trabeculoplasty (SLT)

SUMMARY:
Examination and follow-up of efficacy and safety of SLT in patients with unsufficient IOP control despite maximum tolerated topical therapy. In addition, it will be examined whether medical treatment can be reduced after the SLT procedure and whether filtering surgery - as the only remaining option - may be postponed.

DETAILED DESCRIPTION:
SLT (Selective Laser Trabeculoplasty) uses the Nd:YAG-Lasers (wavelength 532nm, Q-switched, frequency-doubled). Thanks to the low laser energy used and the short duration of treatment, only pigmented cells of the trabecular meshwork are targeted and selectively treated. Neighboring, non-pigmented cells and tissue are spared collateral and thermic damage, the architecture of the trabecular meshwork remains intact. The SLT procedure uses less than 1% of the energy of the ALT procedure with an extremely low pulsation duration.

Several studies confirm the effective IOD reduction of SLT and rate the procedure as an relatively safe and effective therapy for glaucoma. Also repeated use of the SLT procedure is considered as meaningful. Meanwhile the SLT procedure is used as primary and supplementary treatment of glaucoma and study confirmed that the SLT procedure was just as effective as administration of Latanoprost in reducing IOD in newly-diagnosed glaucoma.

ELIGIBILITY:
Inclusion criteria: Patients with

* primary open angle glaucoma (including normal tension glaucoma)
* pseudoexfoliation glaucoma
* pigment dispersion glaucoma

Exclusion criteria: previous intraocular surgery closed angle glaucoma pediatric glaucoma inflammatory or uveitic glaucoma unclear view of the trabecular meshwork

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Study Completion 2009-07

PRIMARY OUTCOMES:
IOP lowering effect of SLT in a special patient group | 1 day, 1 , 3, 6 , 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland